CLINICAL TRIAL: NCT00547690
Title: Electro-acupuncture and Strengthening Exercise for Hemiplegic Elbow and Wrist Joints
Brief Title: Acupuncture in Stroke Rehabilitation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Expired IRB approval
Sponsor: Wen Liu, Ph.D. (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor-Investigator, Wen Liu, Ph.D., Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 9179; 0555637Z
Record Dates: First submitted 2007-10-18; First posted 2007-10-22 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Acupuncture and strength training
  Interventions: Other: Acupuncture and Strengthening
- 2 (Other): Strength training
  Interventions: Other: Strengthening Alone

INTERVENTIONS:
Other: Acupuncture and Strengthening — Acupuncture and strengthening
  Arms: 1
Other: Strengthening Alone — Strengthening training program
  Arms: 2

SUMMARY:
The primary purpose of the study is to examine the effect of acupuncture treatment when combined with strength training on the motor functional recovery of stroke survivors

DETAILED DESCRIPTION:
In this study, we compare the effect on motor functional improvement between a combined acupuncture and strength training program and the strength training alone. The results may allow us to determine whether the acupuncture may bring in additional benefit to the motor recovery in the upper limb in stroke survivors

ELIGIBILITY:
Inclusion Criteria:

* After stroke (>6 months)

Exclusion Criteria:

* Other neurological diseases

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2003-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Motor Scores | Before and After 6 Week Treatment

SECONDARY OUTCOMES:
Active wrist ROM | Before and After 6 Week Treatment
Quantitative Measure of Muscle Spasticity | Before and After 6 Week Treatment
Ashworth Score | Before and After 6 Week Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wen Liu, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States